CLINICAL TRIAL: NCT00216177
Title: Randomised, Multicenter, Open-label, Parallel-group Study Comparing Adalimumab 40 mg s.c. Eow Versus Infliximab 3 mg/kg i.v. Every 6 Weeks in Rheumatoid Arthritis Patients With Unsustainable Clinical Response to Infliximab 3 mg/kg Every 8 Weeks
Brief Title: Comparison of Adalimumab and Infliximab Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Henrik Skjodt, Hvidovre Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 232-003; EudraCT no: 2005-001633-14; Switch/HUM 05-001
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Infliximab — Remicade
  Other Names: remicade
Drug: Adalimumab — Humira
  Other Names: Humira

SUMMARY:
The purpose of this study is to establish whether RA patients with moderate to severe disease activity with unsustainable response to infliximab 3 mg/kg every 8 weeks have better efficacy with adalimumab 40 mg s.c. eow compared to infliximab 3 mg/kg i.v. every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria fulfilled,DAS28-3(CRP > 3.2
* > 6 months prior treatment with infliximab 3 mg/kg i.v. every 8 week with initial response
* Fading clinical response to infliximab
* Negative pregnancy test (women with childbearing potential)
* Use of reliable method of contraception (women with childbearing potential)
* Informed consent

Exclusion Criteria:

* Age less than 18 years
* Lack of co-operability
* Positive serology for hepatitis B or C
* History of positive HIV status
* History of TB or untreated latent TB
* Histoplasmosis or Listeriosis
* Pregnancy or breastfeeding
* Persistent or recurrent infections
* History of cancer
* Uncontrolled diabetes
* Ischaemic heart disease
* Congestive heart failure (NYHA 3-4)
* Active inflammatory bowel disease
* Recent stroke (within 3 months)
* History of or current inflammatory joint disease other than RA
* Previous diagnosis or signs of central nervous system demyelinating disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-01 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving combined good or moderate EULAR responses at week 24 | six months

SECONDARY OUTCOMES:
ACR20/50/70 response at week 2, 6, 12, 18 and 24 | six months

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Skjodt, MD, PhD, Principal Investigator — Hvidovre University Hospital
Locations (6):
- Denmark (6):
  - Hvidovre Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Amtssygehus, Copenhagen
  - Glostrup Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Graasten Gigthospital, Gråsten